CLINICAL TRIAL: NCT01119924
Title: Phase IV Study for Evaluation the Efficacy and Safety of Mirtazapine (Smilon) in Depression Patients With Pain
Brief Title: A Clinical Study for Assessment of the Efficacy and Safety of Mirtazapine (Smilon) in Depression Patients With Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Collaborators: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Hsu Cindy, Nang Kuang Pharmaceutical Co., LTD
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB098-33
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Depression; Pain
Keywords: Mirtazapine; Smilon; Depression; Pain
MeSH Terms: conditions — Depression; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirtazapine (Active Comparator): Mirtazapine 15mg/day or placebo once a day on the fist week, then 30 mg/day or placebo once a day, and then for 7 consecutive weeks
  Interventions: Drug: Smilon®
- Placebo (Placebo Comparator): Smilon® tablet 15mg mg/day or placebo, once a day on the first week, and then for 7 consecutive weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Smilon® — Smilon® tablet 15mg mg/day or placebo, once a day on the first week, and then for 7 consecutive weeks
  Arms: Mirtazapine
Drug: Placebo — Smilon® tablet 15mg mg/day or placebo, once a day on the first week, and then for 7 consecutive weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of Smilon® in the Depression Patients with pain. Eligible patients will be randomly assigned to 1 of 2 arms, either Smilon® or placebo, and will receive the treatment for 8 weeks in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 20-65 years
* Diagnosis of at least one chronic pain syndrome and the diagnosis of concomitant depression according to DSM-IV criteria
* Have a mean weekly pain score of at least 30 mm on the 100-mm visual analog scale (VAS) of the Short-Form McGill Pain Questionnaire (SF-MPQ) before study entry

Exclusion Criteria:

* Women of child bearing potential who are pregnant, breastfeeding or not using effective contraceptives
* Known hypersensitivity to Mirtazapine or any of its components
* Subjects who have a clinically significant or unstable medical or psychiatric condition
* Subjects who have received nerve blocks or acupuncture for pain relief

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain intensity using the visual analog scale (VAS) | 8-week treatment

SECONDARY OUTCOMES:
Evaluation of Severity of depressive symptom using the Depression and Somatic Symptoms Scale (DSSS) | 8-week treatment
Evaluation of Severity of depressive and anxious symptom using the Hamilton depression scale (HAM-D) and Hamilton anxiety scale (HAM-A) | 8-week treatment
Evaluation of quality of life assessed by a 28-item WHOQoL self-administered questionnaire | 8-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tsai Hsin Chi, Principal Investigator — Buddhist Tzu Chi General Hospitsl
Locations (1):
- Nang Kuang Pharmaceutical Co., LTD, Tainan, Xinhua Township, Taiwan